CLINICAL TRIAL: NCT00366834
Title: A Phase III, Multicenter, Randomized, Double-Blind, Active Controlled, Parallel Group Study of the Safety and Efficacy of the Intravenous and Oral Formulations of the Neurokinin-1 Receptor Antagonist Casopitant (GW679769) in Combination With Ondansetron and Dexamethasone for the Prevention of Nausea
Brief Title: Intravenous And Oral Casopitant (GW679769) For The Prevention Of Chemotherapy Induced Nausea And Vomiting
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NKV102549
Record Dates: First submitted 2006-08-17; First posted 2006-08-21 (Estimated); Last update posted 2012-09-10 (Estimated); Status verified 2012-06

CONDITIONS: Vomiting; Nausea; Nausea and Vomiting, Chemotherapy-Induced
Keywords: Anthracycline; Cyclophosphamide; Moderately; Nausea; Emetogenic; Vomiting
MeSH Terms: conditions — Vomiting; Nausea | interventions — casopitant; Ondansetron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Control (Placebo Comparator): ondansetron 8 mg oral twice daily on Day 1-3 and dexamethasone 8 mg IV on Day 1 + placebo
  Interventions: Drug: Dexamethasone intravenous; Drug: Ondansetron oral tablets; Drug: placebo
- Single dose oral (Experimental): ondansetron 8 mg oral twice daily on Day 1-3 and dexamethasone 8 mg IV + casopitant 150 mg on Day 1
  Interventions: Drug: Casopitant (GW679769) oral tablets; Drug: Dexamethasone intravenous; Drug: Ondansetron oral tablets
- 3-day oral (Experimental): ondansetron 8 mg oral twice daily on Day 1-3 and dexamethasone 8 mg IV + casopitant 150 mg on Day 1 + 50 mg on days 2 & 3
  Interventions: Drug: Casopitant (GW679769) oral tablets; Drug: Dexamethasone intravenous; Drug: Ondansetron oral tablets
- 3-day IV/oral (Experimental): ondansetron 8 mg oral twice daily on Day 1-3 and dexamethasone 8 mg IV on Day 1 + 90 mg IV casopitant on day 1 and 50 mg oral casopitant on days 2 & 3
  Interventions: Drug: Casopitant (GW679769) oral tablets; Drug: Casopitant (GW679769) intravenous; Drug: Dexamethasone intravenous; Drug: Ondansetron oral tablets

INTERVENTIONS:
Drug: Casopitant (GW679769) oral tablets
  Arms: 3-day IV/oral; 3-day oral; Single dose oral
Drug: Casopitant (GW679769) intravenous
  Arms: 3-day IV/oral
Drug: Dexamethasone intravenous
Drug: Ondansetron oral tablets
  Other Names: Dexamethasone intravenous; Casopitant (GW679769) oral tablets; Casopitant (GW679769) intravenous
Drug: placebo — casopitant placebo
  Arms: Control

SUMMARY:
This is a Phase III trial designed to demonstrate that casopitant (GW679769) plus dexamethasone and ondansetron is more effective in the prevention of vomiting than dexamethasone and ondansetron alone following the administration of moderately emetogenic chemotherapy.

DETAILED DESCRIPTION:
A Phase III, Multicenter, Randomized, Double-Blind, Active Controlled, Parallel Group Study of the Safety and Efficacy of the Intravenous and Oral Formulations of the Neurokinin-1 Receptor Antagonist, Casopitant (GW679769) in Combination with Ondansetron and Dexamethasone for the Prevention of Nausea and Vomiting Induced by Moderately Emetogenic Chemotherapy

ELIGIBILITY:
Inclusion criteria:

* A subject will be considered eligible for inclusion in this study only if all of the following criteria apply:
* Subject understands the nature and purpose of this study and the study procedures and has signed an informed consent form for this study to indicate this understanding.
* At least 18 years of age.
* Is scheduled to receive their first course of an anthracycline and cyclophosphamide containing moderately emetogenic chemotherapy regimen for the treatment of a solid malignant tumor as outlined in Section 8.1.1.
* Has an ECOG performance status of 0, 1, or 2.
* Hematologic and metabolic status must be adequate for receiving a moderately emetogenic regimen and meet the following criteria:

  * Total Neutrophils ≥ 1500/mm³(Standard units : ≥1.5 x 10^9/L)
  * Platelets ≥ 100,000/mm³ (Standard units: ≥100.0 x 10^9/L)
  * Bilirubin ≤ 1.5 x ULN
  * Liver enzymes must be below the following limits:

    * Without known liver metastases: Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) ≤ 2.5 x upper limit of normal.
    * With known liver metastases: AST and/or ALT ≤ 5.0 x upper limit of normal.
* Is willing and able to complete daily components of the subject diary for each study cycle.
* Women of childbearing potential; must commit to consistent and correct use of an acceptable method of birth control; GSK acceptable contraceptive methods, when used consistently and in accordance with both the product label and the instructions of a physician, are as follows:

  1. Non-childbearing potential (i.e., physiologically incapable of becoming pregnant, including any female who is post-menopausal. For purposes of this study, postmenopausal is defined as one year without menses)
  2. child-bearing potential: must have a negative serum pregnancy test result or negative urine dipstick pregnancy test within 24 hours prior to the first dose of investigational product of Cycle 1, Day 1 and agrees to one of the following:

     * male partner who is sterile prior to the female subject's entry into the study and is the sole sexual partner for that female subject
     * oral contraceptives (e.g., oral, injectable, or implantable) with double-barrier method of contraception consisting of spermicide with either condom or diaphragm for a period after the trial to account for potential drug interaction (minimum of six weeks)
     * double-barrier method of contraception consisting of spermicide with either condom or diaphragm
     * intra-uterine device (IUD) with a documented failure rate of less than 1% per year
     * complete abstinence from intercourse for two weeks before exposure to the investigational product throughout the clinical trial, and for a period after the trial to account for elimination of the drug (minimum of three days),
     * if subjects indicate they will remain abstinent during the period described above, they must agree to follow GSK guidelines for the consistent and correct use of an acceptable method of birth control should they become sexually active.

Exclusion criteria:

* Has previously received cytotoxic chemotherapy. A history of previous biological or hormonal therapy will be permitted.
* Is a female subject who is pregnant or lactating.
* Has received radiation therapy to the brain, abdomen, or pelvis in the ten days prior to the first dose of study medication or casopitant investigational product and/or will receive radiation therapy to the brain, abdomen, or the pelvis in the six days following the first dose of study medication (ZOFRAN and dexamethasone) or casopitant investigational product.
* Is scheduled to receive taxane therapy during cycle 1. Note that subjects will be permitted to receive taxane therapy in conjunction with one of the allowed MEC regimens during subsequent cycles.
* Has experienced emesis (i.e., vomiting and/or retching) or clinically significant nausea in the 24 hours preceding the first dose of study medication or casopitant investigational product.
* Has a known central nervous system primary or metastatic malignancy, unless successfully treated with excision or radiation and has been medically stable for at least 1 week prior to receiving the first dose of study medication or casopitant investigational product.
* Has history of documented peptic ulcer disease (via endoscopy or x-ray), active peptic ulcer disease, gastrointestinal obstruction, increased intracranial pressure, hypercalcemia, or any uncontrolled medical condition (other than malignancy) which in the opinion of the Investigator may confound the results of the study, represent another potential etiology for emesis and nausea (other than CINV) or pose an unwarranted risk to the subject.
* Has a known hypersensitivity or contraindication to ZOFRAN, another 5-HT3 receptor antagonist, dexamethasone, or any component of casopitant.
* Has previously received an NK-1 receptor antagonist.
* Received an investigational drug in the previous 30 days or is scheduled to receive any investigational drug other than casopitant during the study period.
* Has taken/received any medication of moderate or high emetogenic potential within the 48 hours prior to the first dose of study medication or casopitant investigational product. Opioid narcotics for cancer pain will be permitted if the subject has been on a stable dose and has not experienced emesis or nausea from the narcotics.
* Has taken/received any medication with known or potential antiemetic activity within the 24-hour period prior to receiving study drug. This includes, but is not limited to:

  * 5-HT3 receptor antagonists (e.g., ondansetron, granisetron, dolasetron, tropisetron, ramosetron). Palonestron is not permitted within 7 days prior to administration of investigational product.
  * benzamide / benzamide derivatives (e.g., metoclopramide, alizapride)
  * benzodiazepines (except if the subject is receiving such medication for sleep or anxiety and has been on a stable dose for at least seven days prior to the first dose of casopitant investigational product; however, lorazepam is prohibited 24 hours prior to receiving study drug regardless of reason for use)
  * phenothiazines (e.g., prochlorperazine, promethazine, fluphenazine, perphenazine, thiethylperazine, chlorpromazine)
  * butyrophenone (e.g., haloperidol, droperidol)
  * corticosteroids (e.g., dexamethasone, methylprednisolone; with the exception of topical steroids for skin disorders, inhaled steroids for respiratory disorders, and prophylactic treatment for taxane therapy during subsequent cycles)
  * anticholinergics (e.g., scopolamine, with the exception of inhaled anticholingerics for respiratory disorders e.g., ipratropium bromide)
  * antihistamines (e.g., cyclizine, hydroxyzine, diphenhydramine), except for prophylactic use for taxane therapy during cycle 2-4
  * domperidone
  * cannabinoids
  * mirtazpine
  * olanzapine
* Has taken/received strong or moderate inhibitors of CYP3A4 and CYP3A5 for a specified period prior to administration of casopitant investigational product (see Section 8.2.1 "Inhibitors of CYP3A4 and CYP3A5")
* Has taken/received inducers of CYP3A4 and CYP3A5 within fourteen days prior to the administration of casopitant investigational product. (see Section 8.2.2 "Inducers of CYP3A4 and CYP3A5")
* Is taking the anti-diabetic agent repaglinide or the diuretic torsemide. Investigators are advised to exercise caution if including patients taking the anti-diabetic agents rosiglitazone or pioglitazone, or antimalarial agents such as chloroquine and amodiaquine, as the metabolite of casopitant is a potential inhibitor of CYP2C8 (See Section 8.2.3 "Substrates for CYP2C8" and Section 8.4 "Necessary Caution with CYP2C8 Substrates").
* Is currently taking or plans to take the any of the following CYP3A4 substrates: astemizole, cisapride, pimozide, terfenadine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1840 (Actual)
Dates: Start 2006-07; Primary Completion 2007-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Complete response as assessed by a visual analogue scale and a subject diary over the 120 hours following the first cycle of chemotherapy. | 120 Hours

SECONDARY OUTCOMES:
Complete response over 120 hours following subsequent chemotherapy cycles Use of rescue medication over 120 hours following all chemotherapy cycles Impact on daily life activities over 120 hours, assessed using a subject diary questionnaire | 120 Hours
The proportion of subjects who achieve a complete response during the acute (0-24 hours) and the delayed (24-120 hours) phase following the first cycle of MEC. | approx. 18 mos
The proportion of subjects who achieve a complete response over the first 120 hours, during the acute (0-24 hours), the delayed (24-120 hours), and the overall (0-120 hours) phase following subsequent cycles of MEC. | approx. 18 mos
Maximum nausea score (to assess the severity of nausea), as assessed by a Visual Analogue Scale (VAS) over the first 120 hours and in the acute and delayed phases following each cycle of MEC. | approx. 18 mos
Time to first antiemetic rescue medication, defined as the time elapsed from the start of administration of the MEC regimen to the first use of antiemetic rescue medication. | approx. 18 mos
If a subject withdraws prematurely during the first 120 hours, then the time of withdrawal will be considered to be their time to first use of antiemetic rescue medication, and will be censored. | approx. 18 mos
Time to first emetic event, defined as the time elapsed from the start of administration of the MEC regimen to the first emetic episode. If a subject withdraws prematurely during the first 120 hours, | approx. 18 mos
then the time of withdrawal will be considered to be their time to first emetic episode, and will be censored. | approx. 18 mos
The proportion of subjects who receive rescue medication. | approx. 18 mos
The proportion of subjects reporting significant nausea defined as a maximum nausea score greater than or equal to 25 mm on the VAS. | approx. 18 mos
The proportion of subjects reporting nausea defined as a maximum nausea score greater than or equal to 5 mm on the VAS. | approx. 18 mos
The proportion of subjects achieving complete protection, defined as complete responders who had no significant nausea. | approx. 18 mos
The impact on subjects' daily life activities for the first 120 hours following the first cycle of chemotherapy as assessed by the FLIE questionnaire. | approx. 18 mos
Subject satisfaction with the prophylactic antiemetic regimens, and the willingness of subjects to use the same treatment during future chemotherapy, as assessed by the Subject Satisfaction\Willingness Assessment in the Subject Diary. | approx. 18 mos
Nausea as assessed by a categorical scale, over the first 120 hours following MEC administration. | approx. 18 mos
Assessment of the safety and tolerability of casopitant through: routine physical exam, routine clinical laboratory tests, clinical monitoring and adverse events reporting. | approx. 18 mos
The proportion of subjects who vomit/retch. | approx. 18 mos
The proportion of subjects achieving total control, defined as complete responders who had no nausea. | approx. 18 mos

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (201):
- United States (81):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Glendale, Arizona
  - GSK Investigational Site, Fayetteville, Arkansas
  - GSK Investigational Site, Hot Springs, Arkansas
  - GSK Investigational Site, Jonesboro, Arkansas
  - GSK Investigational Site, Concord, California
  - GSK Investigational Site, Fountain Valley, California
  - GSK Investigational Site, Fresno, California
  - GSK Investigational Site, Greenbrae, California
  - GSK Investigational Site, La Verne, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Orange, California
  - GSK Investigational Site, Poway, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Soquel, California
  - GSK Investigational Site, Norwich, Connecticut
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Boynton Beach, Florida
  - GSK Investigational Site, Brooksville, Florida
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Inverness, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, New Port Richey, Florida
  - GSK Investigational Site, Tamarac, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Augusta, Georgia
  - GSK Investigational Site, Columbus, Georgia
  - GSK Investigational Site, Lawrenceville, Georgia
  - GSK Investigational Site, Centralia, Illinois
  - GSK Investigational Site, Galesburg, Illinois
  - GSK Investigational Site, Skokie, Illinois
  - GSK Investigational Site, Evansville, Indiana
  - GSK Investigational Site, Muncie, Indiana
  - GSK Investigational Site, Terre Haute, Indiana
  - GSK Investigational Site, Mason City, Iowa
  - GSK Investigational Site, Hazard, Kentucky
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Alexandria, Louisiana
  - GSK Investigational Site, Baton Rouge, Louisiana
  - GSK Investigational Site, Metairie, Louisiana
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Pittsfield, Massachusetts
  - GSK Investigational Site, Worcester, Massachusetts
  - GSK Investigational Site, Clinton Township, Michigan
  - GSK Investigational Site, Free Soil, Michigan
  - GSK Investigational Site, Saint Joseph, Michigan
  - GSK Investigational Site, Troy, Michigan
  - GSK Investigational Site, Hattiesburg, Mississippi
  - GSK Investigational Site, Tupelo, Mississippi
  - GSK Investigational Site, Jefferson City, Missouri
  - GSK Investigational Site, Rolla, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Billings, Montana
  - GSK Investigational Site, Great Falls, Montana
  - GSK Investigational Site, Denville, New Jersey
  - GSK Investigational Site, Newark, New Jersey
  - GSK Investigational Site, Somerville, New Jersey
  - GSK Investigational Site, Sparta, New Jersey
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, Buffalo, New York
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Bismarck, North Dakota
  - GSK Investigational Site, Akron, Ohio
  - GSK Investigational Site, Bethlehem, Pennsylvania
  - GSK Investigational Site, Hershey, Pennsylvania
  - GSK Investigational Site, Sayre, Pennsylvania
  - GSK Investigational Site, Mt. Pleasant, South Carolina
  - GSK Investigational Site, Sumter, South Carolina
  - GSK Investigational Site, Corpus Christi, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Richardson, Texas
  - GSK Investigational Site, Logan, Utah
  - GSK Investigational Site, Ogden, Utah
  - GSK Investigational Site, Burlington, Vermont
  - GSK Investigational Site, Everett, Washington
  - GSK Investigational Site, Spokane, Washington
  - GSK Investigational Site, Tacoma, Washington
  - GSK Investigational Site, Huntington, West Virginia
  - GSK Investigational Site, Madison, Wisconsin
- Argentina (5):
  - GSK Investigational Site, Capital Federal, Buenos Aires
  - GSK Investigational Site, Mendoza, Mendoza Province
  - GSK Investigational Site, Rosario, Santa Fe Province
  - GSK Investigational Site, San Miguel de Tucumán, Tucumán Province
  - GSK Investigational Site, Quilmes
- Austria (4):
  - GSK Investigational Site, Salzburg
  - GSK Investigational Site, Sankt Pölten
  - GSK Investigational Site, Vienna
  - GSK Investigational Site, Vöcklabruck
- Belgium (3):
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Ghent
  - GSK Investigational Site, Ottignies
- Bulgaria (3):
  - GSK Investigational Site, Plovdiv
  - GSK Investigational Site, Shumen
  - GSK Investigational Site, Sofia
- Canada (15):
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Moncton, New Brunswick
  - GSK Investigational Site, St. John's, Newfoundland and Labrador
  - GSK Investigational Site, Oshawa, Ontario
  - GSK Investigational Site, Thunder Bay, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Windsor, Ontario
  - GSK Investigational Site, Charlottetown, Prince Edward Island
  - GSK Investigational Site, Greenfield Park, Quebec
  - GSK Investigational Site, Laval, Quebec
  - GSK Investigational Site, Lévis, Quebec
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Québec, Quebec
  - GSK Investigational Site, Sherbrooke, Quebec
  - GSK Investigational Site, Saskatoon, Saskatchewan
- GSK Investigational Site, Zagreb, Croatia
- Czechia (7):
  - GSK Investigational Site, Brno
  - GSK Investigational Site, Chomutov
  - GSK Investigational Site, Ostrava - Poruba
  - GSK Investigational Site, Pardubice
  - GSK Investigational Site, Prague
  - GSK Investigational Site, Tábor
  - GSK Investigational Site, Ústí nad Labem
- Denmark (2):
  - GSK Investigational Site, Herlev
  - GSK Investigational Site, Hilleroed
- Estonia (2):
  - GSK Investigational Site, Tallinn
  - GSK Investigational Site, Tartu
- Germany (10):
  - GSK Investigational Site, Heidelberg, Baden-Wurttemberg
  - GSK Investigational Site, Ingolstadt, Bavaria
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Würzburg, Bavaria
  - GSK Investigational Site, Hamburg, Hamburg
  - GSK Investigational Site, Kassel, Hesse
  - GSK Investigational Site, Würselen, North Rhine-Westphalia
  - GSK Investigational Site, Berlin, State of Berlin
  - GSK Investigational Site, Bad Berka, Thuringia
  - GSK Investigational Site, Jena, Thuringia
- Greece (4):
  - GSK Investigational Site, Athens
  - GSK Investigational Site, Kavala
  - GSK Investigational Site, Pátrai
  - GSK Investigational Site, Thessaloniki
- Hong Kong (4):
  - GSK Investigational Site, Hong Kong
  - GSK Investigational Site, Shatin
  - GSK Investigational Site, Tuenmen
  - GSK Investigational Site, Wan Chai
- Hungary (3):
  - GSK Investigational Site, Győr
  - GSK Investigational Site, Gyula
  - GSK Investigational Site, Veszprém
- GSK Investigational Site, Pune, India
- Ireland (3):
  - GSK Investigational Site, Dublin
  - GSK Investigational Site, Tallaght, Dublin
  - GSK Investigational Site, Wilton, Cork
- Italy (6):
  - GSK Investigational Site, Benevento, Campania
  - GSK Investigational Site, Rome, Lazio
  - GSK Investigational Site, Genoa, Liguria
  - GSK Investigational Site, Sanremo (IM), Liguria
  - GSK Investigational Site, Sassari, Sardinia
  - GSK Investigational Site, Perugia, Umbria
- Latvia (2):
  - GSK Investigational Site, Liepāja
  - GSK Investigational Site, Riga
- Lithuania (3):
  - GSK Investigational Site, Kaunas
  - GSK Investigational Site, Klaipėda
  - GSK Investigational Site, Vilnius
- Mexico (2):
  - GSK Investigational Site, Durango, Durango
  - GSK Investigational Site, Mérida, Yucatán
- GSK Investigational Site, Lahore, Pakistan
- Peru (2):
  - GSK Investigational Site, Lima, Lima Province
  - GSK Investigational Site, Callao
- Philippines (4):
  - GSK Investigational Site, Cebu
  - GSK Investigational Site, Manila
  - GSK Investigational Site, Quezon City
  - GSK Investigational Site, Santa Cruz, Manila
- GSK Investigational Site, Krakow, Poland
- Russia (5):
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Moscow Region
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Samara
  - GSK Investigational Site, Yaroslavl
- Slovakia (4):
  - GSK Investigational Site, Bratislava
  - GSK Investigational Site, Nitra
  - GSK Investigational Site, Poprad
  - GSK Investigational Site, Žilina
- South Africa (6):
  - GSK Investigational Site, Athlone Park, Amanzimtoti
  - GSK Investigational Site, Bloemfontein
  - GSK Investigational Site, Observatory
  - GSK Investigational Site, Panorama
  - GSK Investigational Site, Parktown
  - GSK Investigational Site, Saxonwold, Johannesburg
- GSK Investigational Site, Seoul, South Korea
- Spain (6):
  - GSK Investigational Site, Donostia / San Sebastian
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Ourense
  - GSK Investigational Site, Santiago de Compostela
  - GSK Investigational Site, Segovia
  - GSK Investigational Site, Zamora
- Taiwan (3):
  - GSK Investigational Site, Kaohsiung City
  - GSK Investigational Site, Tainan
  - GSK Investigational Site, Taipei
- GSK Investigational Site, Bangkok, Thailand
- United Kingdom (6):
  - GSK Investigational Site, Chelmsford, Essex
  - GSK Investigational Site, Aberdeen
  - GSK Investigational Site, London
  - GSK Investigational Site, Maidstone
  - GSK Investigational Site, Nottingham
  - GSK Investigational Site, Shrewsbury

REFERENCES:
- [Result] Herrstedt J, Apornwirat W, Shaharyar A, Aziz Z, Roila F, Van Belle S, Russo MW, Levin J, Ranganathan S, Guckert M, Grunberg SM. Phase III trial of casopitant, a novel neurokinin-1 receptor antagonist, for the prevention of nausea and vomiting in patients receiving moderately emetogenic chemotherapy. J Clin Oncol. 2009 Nov 10;27(32):5363-9. doi: 10.1200/JCO.2009.21.8511. Epub 2009 Oct 5. PMID 19805683